CLINICAL TRIAL: NCT01866761
Title: Analysis of the Relationship Between Periodontal Disease and Atherosclerosis Within a Local Cooperation System of Japanese Medical Services
Brief Title: Relationship Analysis Between Periodontal Disease and Atherosclerosis in Japanese Medical Cooperation Services
Acronym: RAPA-JMCS
Status: Completed | Type: Observational
Sponsor: Okayama University (Other)
Responsible Party: Principal Investigator, Shogo Takashiba, DDS, PhD, Professor of Periodontal Science, Professor, Okayama University
Other Study IDs: TCHK_OU-RN605
Record Dates: First submitted 2013-05-20; First posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Periodontal Disease; Atherosclerosis
MeSH Terms: conditions — Periodontal Diseases; Atherosclerosis | interventions — Periodontal Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Periodontitis, Lifestyle-related disease
  Interventions: Procedure: Periodontal treatment

INTERVENTIONS:
Procedure: Periodontal treatment

SUMMARY:
Objective: We aimed at analyzing the relationship between periodontal disease and atherosclerosis in medical treatment and periodontal treatment under medical and dental care across borders in a local cooperation system of Japanese medical services.

Materials and methods:

* A prospective multi-center case cohort study was conducted on 37 ambulatory medical patients (with lifestyle-related diseases under consultation in either of the medical clinics registered as collaborative investigation facilities) and 79 periodontal patients (who were seen by the dental clinics registered as collaborative investigation facilities).
* Medical treatment and clinical periodontal treatment were provided on the subjects under medical and dental care across borders by each internal medicine and dental clinics.
* Systemic examination of lifestyle-related disease and periodontal examination were performed before and after periodontal treatment, and the relationships between periodontal and atherosclerosis-related clinical markers were analyzed before and after periodontal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal disease: inflamed gingiva with positive for bleeding on probing or teeth with probing pocket depth more than 4 mm Lifestyle-related disease: Plaques are included when maximum IMT is measured. Furthermore, hypertension was defined as systolic blood pressure of more than 140 mm Hg or diastolic pressure of more than 90 mm Hg, or both, or patients already being treated by anti-hypertensive agents. Hypercholesterolemia was defined by serum concentration of LDL-C of more than 140 mg/dL, or patients already being treated by lipid-lowering agents. Diabetes mellitus was defined by HbA1c of more than 6.9 % (NGSP value) or fasting blood sugar of more than 126 mg/dl or both, or patients already being treated by agents for diabetes.

Exclusion Criteria:

* At initial consultation and examination (Baseline), patients with less than 6 months after the onset of acute myocardial infarction (AMI), and with a past history or complication of serious heart disease were excluded. Similarly, those with less than 6 months after cardiovascular revascularization surgery, less than 6 months after the onset of cerebrovascular disorder, or serious liver disease or renal disease were also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This clinical study was performed by the local clinics which belonged to Tokyo Medical Practitioners Association, Tokyo Dental Practitioners Association, and Chiba Medical Practitioners Association. 37 patients (with lifestyle-related diseases under consultation in either of 16 medical clinics), and 79 periodontal patients (not undergoing treatment at a medical clinic,) were enrolled. The subjects constituted a broad cross-section of the local society. Medical treatment at an internal medicine clinic and clinical periodontal treatment including periodontal surgery at a dental clinic were performed on all the subjects. Twenty-six patients dropped out of the study and medical treatment and periodontal treatment were provided to the remaining 90 subjects (mean ages: 59.2 ± 12.3 yrs).
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2008-11; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Relation between probing pocket depth and anti-periodontopathic bacteria IgG antibody titer for periodontitis and the MAX intima-media thickness, urea sugar, urea protein, urea occult blood, creatinine, and eGFR for atherosclerosis | an expected average of 1.5 year
  At following 3-time points; Baseline, After initial preparation of periodontal treatment, Starting point of supportive periodontal therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Okayama University of Graduate School of Medicine, Dentistry and Pharmaceutical Sciences, Okayama, Okayama-ken, Japan